CLINICAL TRIAL: NCT03701620
Title: Heart Rate Variability in Children With Traumatic Brain Injury and Neurological Outcome
Brief Title: Heart Rate Variability in Children With Traumatic Brain Injury
Acronym: HRV-TBI
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Laurence Ducharme-Crevier, Pediatric intensivist, Principal Investigator, St. Justine's Hospital
Other Study IDs: HSJ 2018-1575
Record Dates: First submitted 2018-10-03; First posted 2018-10-10 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Brain Injury; Child Development
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HRV monitoring — HRV monitoring derived from electrocardiogram

SUMMARY:
Using a prospective cohort of children admitted to the PICU, the investigators will determine HRV monitoring is feasible, if a decreased HRV in the 7 days following moderate or severe TBI in children is associated with a worse outcome 6 months post-TBI and investigate HRV as a tool that can predict adverse events (neurological crisis) within 2 days following TBI.

DETAILED DESCRIPTION:
This is a single center prospective cohort study of 15 children <18 years, admitted to the PICU at the CHU Sainte-Justine (CHUSJ) with moderate or severe TBI (<24 hours). Neurodevelopment outcome of children will be evaluated 6 months post TBI.

ELIGIBILITY:
Inclusion Criteria:

* <18 years
* admitted to the PICU at the CHUSJ
* moderate TBI (Glasgow Coma Scale (GCS): 9-12) or severe TBI (GCS ≤8) as - - assessed 30 minutes after TBI or upon arrival in the emergency room
* written parental consent.

Exclusion Criteria:

* children fulfilling brain death criteria at the time of PICU admission (GCS 3 and loss of all brain stem reflexes)
* children with a pacemaker or with previously diagnosed arrhythmia (HRV monitoring not reliable)
* inflicted trauma (different underlying pathophysiology)
* patients or parents who do not speak or read English or French.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children requiring PICU admission after TBI
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
% of the time with reliable HRVmonitoring in children with TBI | 1 year
  Feasibility of having a reliable capture and analysis of HRV 7 days post TBI

SECONDARY OUTCOMES:
Rate of adverse events preceded by a decreased HRV | 1 year
  Adverse events will be defined as increased intracranial pressure, decreased CPP, seizure and cardiac arrest
HRV and neurological outcome | 1.5 year
  The primary outcome of neurological and functional outcome will be assessed by the Pediatric Glasgow Outcome Scale Extended (P-GOSE) 6 months post TBI. P-GOSE is an 8-point ordinal scale (1= best outcome) The score will be classified as favourable (P-GOSE 1 or 2, or decreased of P-GOSE of 1 point post PICU (∆ P-GOSE ≤1) or unfavourable (P-GOSE ≥3 or ∆ P-GOSE ≥2)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided